CLINICAL TRIAL: NCT05831267
Title: Fibrin Glue Versus Titanium Platelet-rich Fibrin as a Sole Filling Material in Lateral Sinus Lifting With Simultaneous Implant Placement (Randomized Controlled Clinical Trial )
Brief Title: Fibrin Glue Versus Titanium Platelet-rich Fibrin in Lateral Sinus Lifting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sinus_lifting_2022
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Sinus Floor Augmentation; Graftless Sinus Elevation
Keywords: Tenting implant; Fibrin glue; T-PRF
MeSH Terms: interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group 1 (Experimental)
  Interventions: Other: Fibrin Glue
- Study group 2 (Experimental)
  Interventions: Other: T-PRF
- Control group (Other)
  Interventions: Other: Negative control

INTERVENTIONS:
Other: Fibrin Glue — Blood samples were collected from the antecubital vein of the right or left arm of the patient and drawn into sterile Titanium tubes immediately. The tubes were then centrifuged for 12 minutes at 2800 rpm and room temperature
  Arms: Study group 1
Other: T-PRF — The contents of the two containers (human fibrinogen, human thrombin) will be mixed with distilled water and then aspirated by two syringes after that, the two solutions will be mixed together and injected into the empty compartment around the dental implant under the sinus mucosal lining using auto mixing applicator.
  Arms: Study group 2
Other: Negative control — this group will not receive any material.
  Arms: Control group

SUMMARY:
Graftless sinus lift with simultaneous implant placement is one of the new techniques, this new technique is presented based on the physiology of intrasinus bone repair.

Schneiderian membrane is known to have an osteogenic nature, now blood clot can be considered autologous osteogenic graft material, to which osteoprogenitors can migrate, differentiate, and regenerate bone.

The aim of this study is to evaluate the effectiveness of using Fibrin glue versus Titanium platelet rich fibrin (T-PRF) as a sole filling material in lateral sinus lifting using with simultaneous implant placement in comparison to a negative control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring implant placement in the posterior maxilla.
* Tooth extractions at the implant sites were performed at least 4 months before surgery.
* Residual bone height between the alveolar bone crest and the sinus floor is 3-5 mm

Exclusion Criteria:

* Maxillary sinus pathologies (sinusitis, long-standing nasal obstruction).
* Any disease-contraindicating surgery (e.g. uncontrolled diabetes).
* Heavy smokers (smoke greater than or equal 25 cigarettes daily).
* Acute oral infections.
* Untreated periodontal disease (gingival index 2 and 3).
* Poor oral hygiene ( Silness-Löe index (score 2-3) ).
* A history of radiotherapy or chemotherapy of the head and neck region.
* Pregnancy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
change in implant stability | Baseline and 6 months
  implant stability will be measures using Ostell device.
change in bone density | Baseline and 6 months
  bone density will be measured using CBCT
change in vertical bone height | Baseline and 6 months
  vertical bone height will be measured using CBCT

SECONDARY OUTCOMES:
change in pain intensity | Through 1 week postopertaive
  This will be assessed using a 10-point Visual Analogue Scale (VAS) in the 1st week postoperatively.
  (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Change in edema score | Through 1 week postopertaive
  The score will be as follows:
  * None (no inflammation)
  * Mild (intraoral swelling confined to the surgical field)
  * Moderate (extraoral swelling in the surgical zone)
  * Severe (extraoral swelling spreading beyond the surgical zone)

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt